CLINICAL TRIAL: NCT01987258
Title: The Acute Effect of Interval-walking
Acronym: acute IWS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Inge Holm, Administrator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-3-2012-141
Record Dates: First submitted 2013-06-28; First posted 2013-11-19 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Glycemic control; excess post-exercise oxygen consumption
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): No exercise (control experiment)
- Interval Walking (Experimental): A one hour interval walking exercise bout
  Interventions: Behavioral: Interval Walking
- Continuous walking (Experimental): A one hour continuous walking exercise bout
  Interventions: Behavioral: Continuous walking

INTERVENTIONS:
Behavioral: Interval Walking
  Other Names: Interval exercise; Interval training
  Arms: Interval Walking
Behavioral: Continuous walking
  Other Names: Continuous exercise; Continuous training
  Arms: Continuous walking

SUMMARY:
Four months of interval walking training (IWT) is superior to energy-expenditure matched continuous walking training (CWT) with regards to weight loss and improvements in glycemic control. The reason for this is unclear. One potential explanation for the differential outcome in weight loss is excess post-exercise oxygen consumption (EPOC), which is defined as the elevated oxygen consumption measured during the hours following an exercise bout. A large EPOC means greater energy expenditure which, if energy intake does not change, leads to a greater weight loss. This weight loss may subsequently improve glycemic control

* Aim 1: To assess the effect of an acute bout of IWT vs. an acute bout of CWT on glycemic control in type 2 diabetics and to assess mechanisms responsible for differences (if any). It is hypothesised that IWT will be more advantageous for improving glycemic control.
* Aim 2: To examine the effect of an acute bout of IWT vs. an acute bout of CWT on EPOC. It is hypothesised that IWT will produce an EPOC of larger magnitude than CWT.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus, type 2

Exclusion Criteria:

* Smoking
* Pregnancy
* insulin dependence
* Contraindication to physical activity (as judged by medical history and screening)
* Evidence of thyroid, liver, lung, kidney or heart disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Glycemic control | Will be assessed immediately after the intervention using a mixed meal tolerance test (duration: 5 hours) followed by continuous glucose monitoring (duration: 48 hours).
  Glycemic control will be assessed after a one hour specific exercise intervention (control/continuous walking/interval walking) in a controlled setting (a mixed meal tolerance test). Moreover, glycemic control will be assessed during the following 2 days in a free-living environment, using continuous glucose monitoring systems.

SECONDARY OUTCOMES:
Excess post-exercise oxygen consumption (EPOC) | Will be assessed immediately after the intervention using a ventilated hood (duration: 5 hours).
  EPOC will be assessed during the hours following the before-mentioned specific exercise bouts using the indirect calorimetry ventilated hood technique.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Karstoft, MD, Principal Investigator — Centre of Inflammation and Metabolism (CIM), Rigshospitalet, Tagensvej 20, section M7641, DK-2100 Copenhagen, Denmark
Locations (1):
- Centre of Inflammation and Metabolism (CIM), Rigshospitalet, Tagensvej 20, section M7641, Copenhagen, Denmark

REFERENCES:
- [Derived] Karstoft K, Christensen CS, Pedersen BK, Solomon TP. The acute effects of interval- Vs continuous-walking exercise on glycemic control in subjects with type 2 diabetes: a crossover, controlled study. J Clin Endocrinol Metab. 2014 Sep;99(9):3334-42. doi: 10.1210/jc.2014-1837. Epub 2014 Jun 6. PMID 24905068